CLINICAL TRIAL: NCT06782243
Title: Comparison of High and Moderate Intensity Statins in Achieving the Target LDL-C Level After Acute Coronary Syndrome: Randomized Controlled Trial
Brief Title: Comparison of High and Moderate Intensity Statins in Achieving the Target LDL-C Level After Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/013
Record Dates: First submitted 2025-01-09; First posted 2025-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Low-Density Lipoprotein Cholesterol; Cardiovascular Diseases; Drug Therapy, Combination
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Patients are allocated into two groups by blocked randomization (6 blocks ensuring balanced allocation).
Masking Description: Randomized (Blocked randomization)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Statin Group (Active Comparator): Participants in this group will receive moderate-intensity statins (Atorvastatin 20 mg, Rosuvastatin 10 mg). The dosage will be in the tablet form, which will be Dosage Form: Tablet Frequency: Once daily Duration: 3 months
  Interventions: Drug: Moderate-Intensity Statins
- High-Intensity Statin Group (Active Comparator): Participants in this group will receive high-intensity statins. Interventions include Atorvastatin 40 mg, or Rosuvastatin 20 mg which will be taken in tablet form.
  Frequency: Once daily Duration: 3 months
  Interventions: Drug: High-Intensity Statins

INTERVENTIONS:
Drug: Moderate-Intensity Statins — Participants will be administered statins based on moderate intensity. This group will receive oral tablets once daily for 3 months. The intervention includes Atorvastatin 20 mg and rosuvastatin 10 mg.
  Other Names: Lipitor (brand name for Atorvastatin), Crestor (brand name for Rosuvastatin)
  Arms: Moderate-Intensity Statin Group
Drug: High-Intensity Statins — Participants will be administered statins based on high intensity. This group will receive oral tablets once daily for 3 months. The intervention includes Atorvastatin 40 mg and rosuvastatin 20 mg.
  Other Names: Lipitor (brand name for Atorvastatin), Crestor (brand name for Rosuvastatin)
  Arms: High-Intensity Statin Group

SUMMARY:
This study evaluates the effectiveness of high- and moderate-intensity statins in achieving target low-density lipoprotein cholesterol (LDL-C) levels in patients with acute coronary syndrome (ACS). The study aims to determine whether moderate-intensity statins can provide comparable benefits to high-intensity statins, particularly for patients at higher risk of adverse effects from higher doses. The findings may inform treatment decisions and reduce financial and clinical burdens on patients.

DETAILED DESCRIPTION:
Statins are the cornerstone of therapy for reducing cardiovascular events in patients with atherosclerotic cardiovascular disease. Current guidelines recommend high-intensity statins for patients with ACS to lower LDL-C levels by 50% or more. However, emerging evidence suggests that the benefits of lowering LDL-C may be independent of the statin dose and type.

This randomized controlled trial investigates the effectiveness of moderate-intensity statins compared to high-intensity statins in reducing LDL-C levels among local populations. The study also explores whether moderate-intensity statins can mitigate adverse effects, such as myopathy or liver dysfunction, commonly associated with high-intensity statin therapy, particularly in populations with lower baseline LDL-C levels and high statin responsiveness.

Participants will be randomly assigned to receive either high-intensity or moderate-intensity statin therapy. The primary outcome measure is the percentage of participants achieving an LDL-C reduction of ≥50% after three months of treatment. Secondary outcomes include the frequency of adverse effects, adherence to therapy, and changes in liver function tests (LFTs) and creatine phosphokinase (CPK) levels.

The study will contribute to understanding the role of moderate-intensity statins in managing LDL-C levels and guide future clinical practices for patient subgroups at risk of adverse effects from high-intensity therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 25 and 85 years.
* Both males and females.
* Diagnosed with acute coronary syndrome as defined in the operational definitions.

Exclusion Criteria:

* History of adverse reactions to statins (e.g., hypersensitivity, myopathy, acute renal failure).
* Current acute liver disease.
* Pregnant or breastfeeding women.
* Participants already on statin therapy

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Reduction in Low-Density Lipoprotein Cholesterol Level | 3 months after the start of treatment
  The primary outcome is the percentage of participants achieving a reduction of ≥50% in LDL-C levels from baseline after 3 months of treatment with either moderate-intensity or high-intensity statins. LDL-C levels will be measured using lipid profiles obtained at baseline (upon admission) and at the end of the study (3 months post-treatment).

SECONDARY OUTCOMES:
Frequency of Myopathy | Throughout the 3-month treatment duration
  The number of participants who develop myopathy as an adverse effect of statins, determined through clinical symptoms and laboratory tests.
Frequency of Elevated Liver Enzymes | Throughout the 3-month treatment duration
  The number of participants with elevated liver enzyme levels (AST and ALT) as an adverse effect of statin therapy, determined through laboratory tests.
Frequency of Elevated Creatine Phosphokinase (CPK) Levels | Throughout the 3-month
  The number of participants with elevated CPK levels as an adverse effect of statin therapy, determined through laboratory tests.
Severity of Adverse Effects | Throughout the 3-month treatment duration
  The severity of adverse effects, such as myopathy, elevated liver enzymes, and elevated CPK levels, categorized using predefined clinical severity scales.
Compliance with Statin Therapy | At 3 months
  Evaluation of participant adherence to prescribed statin therapy, defined as the proportion of days with medication taken as prescribed over the 3-month period. Compliance will be assessed through patient questionnaires and medication logs.
Reduction in Symptom Severity | Baseline and at 3 months
  Reduction in the severity and frequency of symptoms, such as chest pain and fatigue, associated with acute coronary syndrome (ACS). Symptom severity will be measured using the Visual Analogue Scale (VAS) and patient-reported questionnaires.
  VAS scores for symptom severity:
  1. 1-3 Mild pain
  2. 2-6 Moderate pain
  3. 7-10 Severe pain

OTHER OUTCOMES:
Lipid Profile Changes During Follow-Up | 1 month and 3 months
  Changes in LDL-C levels as measured through laboratory investigations at 1 month and 3 months.
  Unit of Measure:
  LDL-C levels (mg/dL)
Liver Function Test (LFT) Results During Follow-Up | 1 month and 3 months
  Changes in liver enzyme levels (AST and ALT) as measured through laboratory investigations at 1 month and 3 months.
  Unit of Measure:
  LFT levels (U/L)
Creatine Phosphokinase (CPK) Levels During Follow-Up | 1 month and 3 months
  Changes in CPK levels as measured through laboratory investigations at 1 month and 3 months.
  Unit of Measure:
  CPK levels (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shafeeq Mehmood, MBBS, Principal Investigator — Khyber Teaching Hospital; Muhammad Faheem Mehmood, MBBS, Principal Investigator — Khyber Teaching Hospital; Syed Muhammad Shabbir Ali Naqvi, Principal Investigator — Clinical Trial Unit, Khyber Medical University Peshawar
Locations (1):
- MTI-KTH (Medical Teaching Institution-Khyber Teaching Hospital), Peshawar-Pakistan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the study will be made available to other researchers upon reasonable request. The shared data will include de-identified participant data such as baseline demographic details, laboratory results, and follow-up outcomes related to LDL-C levels.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be made available starting six months after the publication of the study results and will remain accessible for a period of five years.
Access Criteria: Access to the data will be granted upon approval of a written proposal outlining the purpose of the data request and intended use. Researchers must provide a signed data access agreement to ensure data confidentiality and compliance with ethical standards.

REFERENCES:
- [Background] Reiner Z. Statins in the primary prevention of cardiovascular disease. Nat Rev Cardiol. 2013 Aug;10(8):453-64. doi: 10.1038/nrcardio.2013.80. Epub 2013 Jun 4. PMID 23736519
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804